CLINICAL TRIAL: NCT03061760
Title: Could Urinary Bladder Hypertrophy Influence on Urge Urine Incontinence Development in Patients After Radical Prostatectomy: A Multi-center Study
Brief Title: Effects of Urinary Bladder Hypertrophy on Urge Urine Incontinence After Radical Prostatectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Tomasz Drewa, Prof. dr hab. n. med., Collegium Medicum w Bydgoszczy
Other Study IDs: CMBydgoszczy
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Prostate Cancer; Urinary Incontinence, Urge; Incontinence; Prostatectomy; Overactive Bladder
Keywords: Prostate cancer; Incontinence; Radical prostatectomy; Urge urinary incontinence
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence, Urge; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1. OAB (-) BOO (-): Patients diagnosed with prostate cancer, undergoing radical prostatectomy, with no overactive bladder (OAB) symptoms and without bladder outlet obstruction (BOO). 'Initial evaluation' before the surgery and follow up - 'Evaluation after 1,3,6,9,12 months'.
  Interventions: Procedure: Radical prostatectomy; Diagnostic Test: Initial evaluation; Diagnostic Test: Evaluation after 1,3,6,9,12 months
- 2. OAB (-) BOO (+): Patients diagnosed with prostate cancer, undergoing radical prostatectomy, with no overactive bladder (OAB) symptoms and with bladder outlet obstruction (BOO). 'Initial evaluation' before the surgery and follow up - 'Evaluation after 1,3,6,9,12 months'.
  Interventions: Procedure: Radical prostatectomy; Diagnostic Test: Initial evaluation; Diagnostic Test: Evaluation after 1,3,6,9,12 months
- 3. OAB (+) BOO (+): Patients diagnosed with prostate cancer, undergoing radical prostatectomy, with overactive bladder (OAB) symptoms and with bladder outlet obstruction (BOO). 'Initial evaluation' before the surgery and follow up - 'Evaluation after 1,3,6,9,12 months'.
  Interventions: Procedure: Radical prostatectomy; Diagnostic Test: Initial evaluation; Diagnostic Test: Evaluation after 1,3,6,9,12 months
- 4.OAB (+) BOO (-): Patients diagnosed with prostate cancer, undergoing radical prostatectomy, with overactive bladder (OAB) symptoms and without bladder outlet obstruction (BOO). 'Initial evaluation' before the surgery and follow up - 'Evaluation after 1,3,6,9,12 months'.
  Interventions: Procedure: Radical prostatectomy; Diagnostic Test: Initial evaluation; Diagnostic Test: Evaluation after 1,3,6,9,12 months
- 5.Control group: Healthy volunteer individuals aged 20-40. 'Initial evaluation' made only once.
  Interventions: Diagnostic Test: Initial evaluation

INTERVENTIONS:
Procedure: Radical prostatectomy — Radical prostatectomy due to prostate cancer.
  Groups: 1. OAB (-) BOO (-); 2. OAB (-) BOO (+); 3. OAB (+) BOO (+); 4.OAB (+) BOO (-)
Diagnostic Test: Initial evaluation — Questioners, Ultrasound, Uroflowmetry
Diagnostic Test: Evaluation after 1,3,6,9,12 months — Questioners, Ultrasound, Uroflowmetry
  Groups: 1. OAB (-) BOO (-); 2. OAB (-) BOO (+); 3. OAB (+) BOO (+); 4.OAB (+) BOO (-)

SUMMARY:
This study is designed to evaluate men before radical prostatectomy for the incidence of Overactive Bladder (OAB), as well as urge urine incontinence (UUI) development after the surgery. Patients will be evaluated for signs of OAB and for signs of Bladder Outlet Obstruction (BOO). Afterwards they will be divided into four observational groups. Follow up period is designed to be 12 months.

DETAILED DESCRIPTION:
Radical prostatectomy remains the standard treatment in case of organ-confined and in selected cases of locally advanced prostate cancer. Radical prostatectomy consists of removing the prostate gland and seminal vesicles, ideally with negative surgical margins.

Most of the patients who present urinary incontinence after radical prostatectomy have stress urinary incontinence. However in some cases the post-surgical urinary incontinence is also due to urgency caused by overactive bladder development defined as urge urinary incontinence. Recent clinical observations suggest that men can also develop overactive bladder after radical prostatectomy.

This study is designed to evaluate men before radical prostatectomy for the incidence of Overactive Bladder (OAB) and it's development after the surgery. Before surgery questionnaire assessment of lower urinary tract symptoms will be performed using International Prostate Symptom Score (IPSS) questionnaire. OAB symptoms will be analyzed using King's questionnaire, as well as using two different OAB symptom score (OABSS) designed by Blavis et al. and Homma et al. Each patient will have transabdominal ultrasonographic evaluation of the prostate and urinary bladder structure. Prostatic dimensions width (W), height (H), length (L) and volume will be recorded. The ultrasonography will be done in urinary bladder filling related to normal desire to void. Urinary bladder wall thickness (BWT) and detrusor muscle thickness (DWT) will be measured in sagittal plane in anterior bladder wall. The mean of three following measurements BWT and DWT will be obtained. The urinary bladder weight (UEBW: Ultrasound Estimated Bladder Weight) will be also estimated. After ultrasonography each patient will undergo uroflowmetry with post-void residual estimation.

On the results above 4 groups will be formed

Group 1 OAB (-) BOO (-)

Group 2 OAB (-) BOO (+)

Group 3 OAB (+) BOO (+)

Group 4 OAB (+) BOO (-)

The investigators will obtain detail information about the surgery (time, blood loss, histopathological outcome, nerve sparing, complications).

After the initial evaluation of the patients before surgery, the control evaluation is set on 1, 3, 6, 9, and 12 month after radical prostatectomy in groups 1-4 to define the lower urinary tract symptoms after radical prostatectomy related to pre-surgical patient clinical feature. During each of the following controls the investigator will not have the access to previously obtained data from the patient.

In addition, healthy volunteers aged 20 to 40 will be assigned as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Adult men over 40 years old with prostate cancer qualified for radical prostatectomy
* Control group formed from 20 healthy men aged 20-40 years old without any urological conditions and no lower urinary tract symptoms (LUTS).

Exclusion Criteria:

* Neoadjuvant (any time before) or adjuvant radiotherapy or brachytherapy (within the follow-up period of 12 months).
* Macroscopic infiltration of the bladder (pT4).
* Neurological deficiencies, such as stroke, spinal cord injury, multiple sclerosis etc. causing inability to have any control of the bladder.
* Urethral strictures.
* Transurethral resection of the prostate or Adenomectomy performed within 12 months prior to Radical Prostatectomy.
* Any form of constant catheterisation (indwelling catheter, clean intermittent catheterisation).

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men with prostate cancer aged over 40 years old (usually 50-75) undergoing radical prostatectomy before the surgery and observed for 12 months.
  Control group formed from healthy volunteers aged 20-40 years.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Increased incidence OAB - Ultrasonography of bladder wall | 12 months
  Measuring the incidence of overactive bladder and urge urinary incontinence development after radical prostatectomy in patients - characterized by increased urinary wall thickness (changes of urinary bladder wall in ultrasound evaluation measured in sagittal section in millimeters).
  Measurement: Bladder wall thickness, Detrusor Muscle thickness on each follow up visit.
Increased incidence OAB - Questioners | 12 months
  Measuring the incidence of symptoms of overactive bladder and urge urinary incontinence development after radical prostatectomy in patients - characterized by changes found in OABSS survey (Questioners).
  Measurement: OABSS survey on each follow up visit.

SECONDARY OUTCOMES:
Continence | 12 months
  Defined as number of pads used per day during the follow up period.
  Measurement: Number of pads, that patient claims he is using per day at the moment of each follow up visit.
Qmax-Uroflowmetry | 12 months.
  The change of Maximal urine flow in the uroflowmetry test is a good predictor of the quality of urination. The change in Qmax will be observed after radical prostatectomy.
  Measurement: Uroflowmetry on each follow up visit.
Bladder volume during normal desire. | 12 months
  This outcome is designed to check whether and to what extent bladder volume (decreased) influences the development of OAB, worsens the continence and affects quality of life (QoL).
  Measurement: Ultrasound measuring bladder capacity during normal desire on each follow up visit.
Quality of life. | 12 months
  This outcome is designed to check how much incontinence and development of OAB affects the quality of life. King's Quality of Life Questioner will be assessed during each follow up visit.
  Measurement: King's Quality of Life Questioner on each follow up visit.
Quality of urination. | 12 months
  This outcome is designed to check how much the surgery affects the quality of urination itself. IPSS questioner will be assessed during each follow up visit.
  Measurement: IPSS on each follow up visit.
Increased incidence OAB - Ultrasonography - Calculated Bladder weight | 12 months
  Measuring the incidence of overactive bladder and urge urinary incontinence development after radical prostatectomy in patients - characterized by calculated bladder weight (changes of calculated bladder weight in grams).
  Measurement: Calculated Bladder weight on each follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz A Drewa, Prof., Principal Investigator — Collegium Medicum w Bydgoszczy

IPD SHARING:
Plan to Share IPD: No
The summary of all the results will be provided on ClinicalTrials.gov . Individual patient data may be provided after individual request to the extant needed for the requesting researcher.